CLINICAL TRIAL: NCT01500330
Title: Randomised Controlled Study on the Effectiveness of Cupping Massage for Home Use in Chronic Neck Pain [Randomisierte Kontrollierte Studie Zur Wirksamkeit Der Schröpfkopfmassage Als Heimanwendung Bei Chronischen Nackenschmerzen]
Brief Title: Home Use of Cupping Massage in Chronic Neck Pain
Acronym: NaSK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Study coordinator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NaSK
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cupping massage (Experimental): 12 weeks home use of cupping massage (delivered by the partner or friend) twice a week for 20 minutes
  Interventions: Procedure: cupping massage
- control group (Active Comparator): progressive muscle relaxation twice a week for 20 minutes
  Interventions: Procedure: Progressive muscle relaxation

INTERVENTIONS:
Procedure: cupping massage — the upper back is covered in massage oil the cupping glass is drawn along the back muscles
  Arms: cupping massage
Procedure: Progressive muscle relaxation — standardized programme on muscle relaxation according to Jacobson
  Arms: control group

SUMMARY:
The purpose of this randomized controlled study is to determine the effectiveness of cupping massage as home use for patients with chronic nonspecific neck pain compared to relaxation exercise.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* mean neck pain intensity 45mm
* neck pain for at least 3 months
* age 18-75
* partner or friend for the application of the massage

Exclusion Criteria:

* specific neck pain due to trauma, neurological disorder, prolapse, operation, cancer
* severe deformity of the spine
* skin disease, allergy on the neck area
* hemophilia, anticoagulation, antiplatelet disorder
* severe psychiatric disorder
* severe comorbidity
* regular intake of opiates and corticosteroids >10mg prednisolon
* pregnancy
* participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | T2 (84 days)
  Pain intensity on a 100mm visual analogue scale

SECONDARY OUTCOMES:
Pain diary | week 12
  Pain intensity on a visual analogue scale
pain intensity in motion | T2 (84 days)
  Pain intensity induced by flexion, extension, lateral flexion and rotation of the head
pain quality | T2 (84 days)
  sensory and affective pain quality, questionnaire
well being | T2 (84 days)
  Well being measured by questionnaire (FEW16)
Quality of life | T2 (84 days)
  measured by the SF-36
Stress perception | T2 (84 days)
  Measured by the PSQ20
Control belief | T2 (84 days)
  measured by the GKÜ (questionnaire on control beliefs)
Pressure pain threshold | T2 (84 days)
  pressure pain threshold measured with an algometer on predefined muscles and the pain maximum
Safety | T2(84 days)
  all adverse events are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rampp, MD, Principal Investigator — Chair of Complementary and Integrative Medicine, University Duisburg-Essen, Germany
Locations (1):
- Klinik für Naturheilkunde, Essen, Germany

REFERENCES:
- [Result] Lauche R, Materdey S, Cramer H, Haller H, Stange R, Dobos G, Rampp T. Effectiveness of home-based cupping massage compared to progressive muscle relaxation in patients with chronic neck pain--a randomized controlled trial. PLoS One. 2013 Jun 7;8(6):e65378. doi: 10.1371/journal.pone.0065378. Print 2013. PMID 23762355
- See also: Homepage "Klinik für Naturheilkunde" — http://www.kliniken-essen-mitte.de/leistung/fachabteilungen/naturheilkunde-u-integrative-medizin/home.html